CLINICAL TRIAL: NCT01138007
Title: Study AK1113351, a Fixed Dose Study of 323U66 SR in the Treatment of Major Depressive Disorder (MDD) - a Multi-center, Placebo-controlled, Randomized, Double-blind, Parallel-comparison Study
Brief Title: A Fixed Dose Study of 323U66 SR in the Treatment of Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 113351
Record Dates: First submitted 2010-06-03; First posted 2010-06-07 (Estimated); Results first posted 2013-05-06 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-06

CONDITIONS: Depressive Disorder, Major
Keywords: Bupropion; 323U66 Sustained Release (SR); MDD (Major Depressive Disorder); IVRS HAM-D; IDS-SR; MADRS
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 323U66 SR 150 mg cohort (Experimental): 323U66 SR 150 mg tablet is orally administered once in the morning and 323U66 SR 150 mg placebo tablet is orally administered once in the evening throughout the treatment phase.
  Interventions: Drug: 323U66 SR 150 mg tablet; Drug: 323U66 SR 150 mg placebo tablet
- 323U66 SR 300 mg cohort (Experimental): 323U66 SR 150 mg tablet is orally administered once in the morning and 323U66 SR 150 mg placebo tablet is orally administered once in the evening during the first week of the treatment phase. At the second week, 323U66 SR 300mg cohort is up-titrated to a daily dose of 323U66 SR 300 mg, administered as 323U66 SR 150 mg tablet twice daily in the morning and in the evening, and the same daily dose is maintained to administer until the end of the treatment phase.
  Interventions: Drug: 323U66 SR 150 mg tablet; Drug: 323U66 SR 150 mg placebo tablet
- Placebo cohort (Placebo Comparator): 323U66 SR placebo tablet is orally administered twice daily throughout the treatment phase.
  Interventions: Drug: 323U66 SR 150 mg placebo tablet

INTERVENTIONS:
Drug: 323U66 SR 150 mg tablet — 323U66 SR 150 mg tablet is orally administered once in the morning and/or once in the evening during the teatment phase.
  Arms: 323U66 SR 150 mg cohort; 323U66 SR 300 mg cohort
Drug: 323U66 SR 150 mg placebo tablet — 323U66 SR 150 mg placebo tablet is orally administered once in the evening and/or once in the morning during the teatment phase.

SUMMARY:
This is a multi-center, placebo-controlled, randomized, double-blind, parallel-comparison study to confirm the efficacy of 323U66 Sustained Release (SR) orally administered to patients with MDD (Major Depressive Disorder) at doses level of 150 mg/day and 300 mg/day for 8 weeks based on the decrease in MADRS (Montgomery-Asberg Depression Rating Scale) total score, and to evaluate the safety based on adverse events, clinical laboratory tests and vital signs.

ELIGIBILITY:
Inclusion Criteria:

[At the start time of the run-in phase]

* Subject must have a primary diagnosis of major depressive disorder as classified by the DSM-IV-TR criteria as below (however, to exclude those accompanied by comorbid psychiatric disorders), and be showing currently a symptom of depression or depressive status: Major depressive disorder, single episode (296.2x); Major depressive disorder, recurrent (296.3x).
* Subject must have a total score of >=20 on the IVRS HAM-D (17 items).
* Subject must have a total score of >=25 on the IDS-SR.
* Subject must have a score of >=1 on 4 out 5 items on the 5-item subscale of the IDS-SR (Item 19, 20, 21, 22 and 30), and a total score of >=7 on the 5-item subscale of the IDS-SR.
* Subject must have a CGI-SI score of >=4 (i.e., Moderately ill or much worse).
* Subject must have the current depressive episode's duration of >=8 weeks but <24 months.
* Subject is outpatient.
* Subject must show QTc <450 millisecond (msec) or <480msec with Bundle Branch Block - values based on either single ECG values or triplicate ECG averaged QTc values obtained over a brief recording period.
* Subject must show a value less than twice of the upper limit of normal value range of AST (GOT) and ALT (GPT), and a value <=1.5 times of the upper limit of normal value range of both Al-P and total bilirubin (however, subject who shows >35% of direct bilirubin with a value >=1.5 times of the upper limit of normal range of total bilirubin regards eligible).
* Subject must read and write at a level sufficient to provide written informed consent prior to study participation and complete study-related materials. If subject is <20 years of age at the time of giving consent, both the subject himself / herself and his / her proxy consenter must give written informed consent.

[At the start time of the treatment phase]

* Subject must have a total score of >=20 of the IVRS-based HAM-D (17 items).
* Subject whose IVRS HAM-D (17 items) total score has not been increased or decreased by >25% during the run-in phase.
* Subject must have a total score of >=25 on the IDS-SR.
* Subject must have a score of >=1 on 4 out 5 items on the 5-item subscale of the IDS-SR (Item 19, 20, 21, 22 and 30), and a total score of >=7 on the 5-item subscale of the IDS-SR.
* Subject must have a CGI-SI score of >=4 (i.e., Moderately ill or much worse).

Exclusion Criteria:

[At the start time of Run-in phase (Visit 1)]

* Subject has predispositions to seizure: who currently has or has a past history of seizure or seizure disorder, more than a single febrile seizure in infancy, cerebral tumour, or head / brain injury (traumatic); who has a family history of idiopathic seizure; who is diabetic patient with treating by oral hypoglycaemics or insulin; who uses drugs lowering the threshold of seizure.
* Subject has a history or current diagnosis of anorexia nervosa (DSM-IV-TR 307.1) or bulimia (DSM-IV-TR 307.51).
* Subject has a primary DSM-IV diagnosis of, or received treatment for, panic disorder, obsessive compulsive disorder (OCD), posttraumatic stress disorder (PTSD), or acute stress disorder within 12 months before the start time of Run-in phase.
* Subject has a DSM-IV diagnosis of schizophrenia, or other psychotic disorder(s) including bipolar disorder.
* Subject has a history of or currently has manic episode(s).
* Subject has any other DSM-IV axis II diagnosis that would suggest non-responsiveness to pharmacotherapy or non-compliance with the protocol (e.g., antisocial, borderline disorder or narcissistic personality disorder).
* Subject starting psychotherapy (except for supportive psychotherapy not aimed at therapeutic efficacy and unlikely to affect efficacy evaluation) or a cognitive behaviour therapy within 12 weeks before start time of the run-in phase.
* Subject received electroconvulsive therapy (ECT) within 24 weeks before start time of the run-in phase.
* Subject took MAO inhibitors (selegiline hydrochloride) within 2 weeks before start time of the run-in phase.
* Subject who has undergone treatment with a depot neuroleptic in the past.
* Subject has systolic blood pressure of >=160 mmHg or diastolic pressure of >=100 mmHg.
* Subject 1) is possibly pregnant, 2) is pregnant, lactating, or 3) does not agree to use contraceptive method(s) specified in the protocol to avoid pregnancy during the study (females only). Or subject wants to become pregnant during the study (females only).
* Subject has a history of alcohol / substance abuse or dependence within 12 months before start time of the run-in phase and/or has a positive result in a urine test for illicit drug use at start time of the run-in phase.
* Subject, who in the opinion of the investigator (or sub-investigator), poses a current serious suicidal risk or has made a suicide attempt within the past 6 months.
* Subject took another investigational product for the NDA filing or for the post manufacturing / marketing approval study within 12 weeks before start time of the run-in phase.
* Subject is currently participating in another clinical study in which the subject is or will be exposed to an investigational or non-investigational drug or medical device.
* Subject has a history of non-responsiveness to 323U66 SR treatment in the investigational clinical trial for major depressive disorder.
* Subject has a history of withdrawal from the investigational clinical trial of 323U66 SR for major depressive disorder due to any adverse event(s).
* Subject has a history of hypersensitivity to 323U66 (bupropion).
* Subject, who in the opinion of the investigator (or sub-investigator), has a risk of homicide.
* Subject has serious cerebral disease(s).
* Subject has serious physical symptom(s) (i.e., cardiac / hepatic / renal / hematopoietic disorder(s)).
* Subject whose major depressive disorder is due to direct physiological effects of a general medical condition(s) (e.g. hypothyroidism, Parkinson's disease, chronic pain).
* Subject is complicated by chronic hepatitis B or C being positive in test of hepatitis B surface antigen (HbsAg) or hepatitis C antibody.
* Subject who is in the process of quitting smoking with nicotine formulation.
* Subject has previously failed adequate (in terms of dose and duration of therapy) courses of pharmacotherapy with at least two different classes of antidepressants.
* Subjects undergoing abrupt discontinuation of alcohol or sedatives.
* Subject is inappropriate for participating in the study that is felt by the investigator (or sub-investigator).

[At the start time of the treatment phase]

* Subject, who in the opinion of the investigator (or sub-investigator), poses a current serious suicidal risk.
* Subject is inappropriate for participating in the study that is felt by the investigator (or sub-investigator).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 572 (Actual)
Dates: Start 2010-06-17; Primary Completion 2012-08-01 (Actual); Study Completion 2012-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (19):
- Japan (16):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Fukushima
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Nara
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saga
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokyo
- South Korea (3):
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 113351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 572 participants were enrolled in the study; however, 3 of these participants were mistakenly registered and were not randomized to study treatment.
Pre-assignment Details: Participants who met the inclusion criteria enrolled in the 1- to 2-week Run-in Phase before entering the 8-week Treatment Phase, followed by the 2-week Follow-up Phase. In the Run-in Phase, the previous/existing prohibited medications administered were washed out, and participants' clinical symptoms were carefully monitored.
Groups:
- Placebo: A 323U66 sustained release (SR) placebo tablet was administered orally twice daily, in the morning and the evening (Dose level 1 and 2), for 8 weeks.
- 323U66 SR 150 mg: A 323U66 SR 150 milligram (mg) tablet was administered orally once in the morning, and a 323U66 SR 150 mg placebo tablet was administered orally once in the evening, with an interval of at least 8 hours between successive doses (Dose level 1 and 2), for 8 weeks.
- 323U66 SR 300 mg: A 323U66 SR 150 mg tablet was administered orally once in the morning, and a 323U66 SR 150 mg placebo tablet was administered orally once in the evening, with an interval of at least 8 hours between successive doses, during the first week of the Treatment Phase (Dose level 1). At Week 2, participants were up-titrated to a daily dose of 323U66 SR 300 mg, administered as a 323U66 SR 150 mg tablet twice daily, in the morning and in the evening, with an interval of at least 8 hours between successive doses (Dose level 2). Dose level 2 was maintained from Week 2 to Week 8.
Period: Overall Study
Arm/Group | Placebo | 323U66 SR 150 mg | 323U66 SR 300 mg
Started | 187 | 190 | 192
Completed | 165 | 160 | 144
Not Completed | 22 | 30 | 48
Not completed — Adverse Event | 4 | 12 | 9
Not completed — Lack of Efficacy | 2 | 0 | 6
Not completed — Protocol Violation | 2 | 3 | 2
Not completed — Protocol-Defined Stopping Criteria | 6 | 1 | 8
Not completed — Lost to Follow-up | 3 | 3 | 5
Not completed — Physician Decision | 0 | 5 | 3
Not completed — Withdrawal by Subject | 5 | 6 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 323U66 SR 150 mg | 323U66 SR 300 mg | Total
Number analyzed (Participants) | 186 | 190 | 188 | 564
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline data were collected in members of the Full Analysis Set (FAS), consisting of all participants who took at least one dose of investigational product and provided at least one efficacy observation at a Treatment Phase visit (i.e., Week 1 or later).
  Years | 37.9 (11.09) | 36.0 (10.42) | 37.5 (10.96) | 37.1 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline data were collected in members of the FAS, consisting of all participants who took at least one dose of investigational product and provided at least one efficacy observation at a Treatment Phase visit (i.e., Week 1 or later).
  Participants
    Female | 101 | 98 | 105 | 304
    Male | 85 | 92 | 83 | 260
Race/Ethnicity, Customized [Number; unit: participants] — Baseline data were collected in members of the FAS, consisting of all participants who took at least one dose of investigational product and provided at least one efficacy observation at a Treatment Phase visit (i.e., Week 1 or later).
  participants
    Asian - Japanese Heritage | 149 | 154 | 147 | 450
    Asian - East Asian Heritage | 37 | 36 | 40 | 113
    Asian - Mixed Race | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at Week 8/Withdrawal
Description: The MADRS scale measures the depression level of a participant. The total score was derived by adding the scores of the following 10 items: 1, Apparent sadness; 2, Reported sadness; 3, Inner tension; 4, Reduced sleep; 5, Reduced appetite; 6, Concentration difficulties; 7, Lassitude; 8, Inability to feel; 9, Pessimistic thoughts; 10, Suicidal thoughts. Each item was scored using a scale of 0 to 6 (a higher score indicates increased severity). The maximum total score is 60; 0, no depression; 60, severely depressed. Change from Baseline in the total score was calculated as the value at Week 8/Withdrawal minus the value at Baseline. The least squared means were estimated based on the Analysis of Covariance (ANCOVA) model including Baseline MADRS score and region as covariates.
Time Frame: Baseline and Week 8/Withdrawal
Population: Full Analysis Set (FAS): all participants who took at least one dose of investigational product and provided at least one efficacy observation at a Treatment Phase visit (i.e. Week 1 or later). Missing values were imputed using Last Observation Carried Forward (LOCF): last observed non-missing value was used to fill missing values at a later point.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | 323U66 SR 150 mg | 323U66 SR 300 mg
Number analyzed (Participants) | 186 | 190 | 188
Scores on a scale | -13.9 (0.77) | -14.4 (0.77) | -12.9 (0.76)
Statistical Analysis 1: Comparison: Placebo vs 323U66 SR 150 mg; Test type: Superiority or Other; p = 0.853, ANCOVA — The p-value was estimated based on the ANCOVA model including Baseline MADRS score and region as covariates. The multiplicity was adjusted by Dunnett's step-down procedure; Least Squared Mean Difference = -0.5, 95% CI 2-sided [-2.7 to 1.7] — The confidence interval was estimated based on the ANCOVA model including Baseline MADRS score and region as covariates
Statistical Analysis 2: Comparison: Placebo vs 323U66 SR 300 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 1.0, Standard Error of Mean 1.00 — In the analysis plan, the second comparison of interest was not to be performed if the first comparison failed to show statistical significance

2. Secondary Outcome: Change From Baseline in the MADRS Total Score at Weeks 1, 2, 4, and 6
Description: The MADRS scale measures the depression level of a participant. The total score was derived by adding the scores of the following 10 items: 1, Apparent sadness; 2, Reported sadness; 3, Inner tension; 4, Reduced sleep; 5, Reduced appetite; 6, Concentration difficulties; 7, Lassitude; 8, Inability to feel; 9, Pessimistic thoughts; 10, Suicidal thoughts. Each item was scored using a scale of 0 to 6 (a higher score indicates increased severity). The maximum total score is 60; 0, no depression; 60, severely depressed. Change from Baseline in the total score was calculated as the value at Week 1, 2, 4 and 6 minus the value at Baseline. The least squared means were estimated based on the ANCOVA model including Baseline MADRS score and region as covariates.
Time Frame: Baseline; Weeks 1, 2, 4, and 6
Population: FAS. Missing values were imputed using LOCF. Only participants who were available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Groups:
- Placebo: A 323U66 SR placebo tablet was administered orally twice daily, in the morning and the evening (Dose level 1 and 2), for 8 weeks.
- 323U66 SR 150 mg: A 323U66 SR 150 mg tablet was administered orally once in the morning, and a 323U66 SR 150 mg placebo tablet was administered orally once in the evening, with an interval of at least 8 hours between successive doses (Dose level 1 and 2), for 8 weeks.
Arm/Group | Placebo | 323U66 SR 150 mg | 323U66 SR 300 mg
Number analyzed (Participants) | 186 | 190 | 188
Scores on a scale
  Week 1, n=182, 187, 184 | -3.4 (0.38) | -2.9 (0.38) | -2.7 (0.38)
  Week 2, n=186, 190, 188 | -6.2 (0.47) | -5.0 (0.47) | -5.0 (0.47)
  Week 4, n=186, 190, 188 | -9.2 (0.61) | -8.3 (0.60) | -8.2 (0.60)
  Week 6, n=186, 190, 188 | -11.8 (0.70) | -11.7 (0.70) | -11.1 (0.69)

3. Secondary Outcome: Change From Baseline in the MADRS Individual Item Scores at Weeks 1, 2, 4, 6, and 8
Description: The MADRS scale measures the depression level of a participant using the following 10 items: 1, Apparent sadness; 2, Reported sadness; 3, Inner tension; 4, Reduced sleep; 5, Reduced appetite; 6, Concentration difficulties; 7, Lassitude; 8, Inability to feel; 9, Pessimistic thoughts; 10, Suicidal thoughts. Each item was scored using a scale of 0 to 6 (a higher score indicates increased severity). Scores for MADRS items 1, 2, 6, 7, and 8 were evaluated for this endpoint. Change from Baseline was calculated as the value at Week 1, 2, 4, 6, and 8 minus the value at Baseline. The least squared means were estimated based on the ANCOVA model including Baseline MADRS score of each item and region as covariates.
Time Frame: Baseline; Week 1, 2, 4, 6, and 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | 323U66 SR 150 mg | 323U66 SR 300 mg
Number analyzed (Participants) | 186 | 190 | 188
Scores on a scale
  Item 1: Week 1, n=182, 187, 184 | -0.5 (0.07) | -0.3 (0.07) | -0.3 (0.07)
  Item 1: Week 2, n=186, 190, 188 | -0.7 (0.08) | -0.5 (0.08) | -0.6 (0.08)
  Item 1: Week 4, n=186, 190, 188 | -1.0 (0.09) | -0.9 (0.09) | -1.0 (0.09)
  Item 1: Week 6, n=186, 190, 188 | -1.4 (0.10) | -1.3 (0.10) | -1.3 (0.10)
  Item 1: Week 8, n=186, 190, 188 | -1.6 (0.10) | -1.6 (0.10) | -1.5 (0.10)
  Item 2: Week 1, n=182, 187, 184 | -0.5 (0.08) | -0.4 (0.08) | -0.5 (0.08)
  Item 2: Week 2, n=186, 190, 188 | -0.8 (0.09) | -0.8 (0.09) | -0.7 (0.09)
  Item 2: Week 4, n=186, 190, 188 | -1.2 (0.10) | -1.2 (0.10) | -1.1 (0.10)
  Item 2: Week 6, n=186, 190, 188 | -1.6 (0.11) | -1.6 (0.11) | -1.4 (0.11)
  Item 2: Week 8, n=186, 190, 188 | -1.8 (0.12) | -2.0 (0.12) | -1.7 (0.12)
  Item 6: Week 1, n=182, 187, 184 | -0.3 (0.07) | -0.4 (0.07) | -0.4 (0.07)
  Item 6: Week 2, n=186, 190, 188 | -0.6 (0.08) | -0.6 (0.08) | -0.7 (0.08)
  Item 6: Week 4, n=186, 190, 188 | -1.0 (0.10) | -1.1 (0.10) | -1.0 (0.09)
  Item 6: Week 6, n=186, 190, 188 | -1.3 (0.10) | -1.4 (0.10) | -1.4 (0.10)
  Item 6: Week 8, n=186, 190, 188 | -1.5 (0.11) | -1.7 (0.11) | -1.6 (0.11)
  Item 7: Week 1, n=182, 187, 184 | -0.3 (0.08) | -0.3 (0.08) | -0.4 (0.08)
  Item 7: Week 2, n=186, 190, 188 | -0.7 (0.09) | -0.6 (0.09) | -0.7 (0.08)
  Item 7: Week 4, n=186, 190, 188 | -1.0 (0.10) | -0.9 (0.10) | -1.1 (0.10)
  Item 7: Week 6, n=186, 190, 188 | -1.4 (0.11) | -1.3 (0.11) | -1.4 (0.11)
  Item 7: Week 8, n=186, 190, 188 | -1.6 (0.11) | -1.6 (0.11) | -1.6 (0.11)
  Item 8: Week 1, n=182, 187, 184 | -0.4 (0.08) | -0.3 (0.08) | -0.3 (0.08)
  Item 8: Week 2, n=186, 190, 188 | -0.8 (0.09) | -0.6 (0.09) | -0.6 (0.08)
  Item 8: Week 4, n=186, 190, 188 | -1.1 (0.10) | -0.9 (0.10) | -1.0 (0.10)
  Item 8: Week 6, n=186, 190, 188 | -1.3 (0.11) | -1.2 (0.11) | -1.3 (0.11)
  Item 8: Week 8, n=186, 190, 188 | -1.7 (0.12) | -1.7 (0.12) | -1.5 (0.11)

4. Secondary Outcome: Number of MADRS Responders at Week 8
Description: The MADRS scale measures the depression level of a participant. The total score was derived by adding the scores of the following 10 items: 1, Apparent sadness; 2, Reported sadness; 3, Inner tension; 4, Reduced sleep; 5, Reduced appetite; 6, Concentration difficulties; 7, Lassitude; 8, Inability to feel; 9, Pessimistic thoughts; 10, Suicidal thoughts. Each item was scored using a scale of 0 to 6 (a higher score indicates increased severity). The maximum total score is 60; 0, no depression; 60, severely depressed. A MADRS responder is defined as a participant with a >=50% reduction from Baseline in the MADRS total score at Week 8.
Time Frame: Baseline and Week 8
Population: FAS. Missing values were imputed using LOCF.
Measure: Number; unit: participants
Arm/Group | Placebo | 323U66 SR 150 mg | 323U66 SR 300 mg
Number analyzed (Participants) | 186 | 190 | 188
participants | 86 | 98 | 82

5. Secondary Outcome: Number of MADRS Remitters at Week 8
Description: The MADRS scale measures the depression level of a participant. The total score was derived by adding the scores of the following 10 items: 1, Apparent sadness; 2, Reported sadness; 3, Inner tension; 4, Reduced sleep; 5, Reduced appetite; 6, Concentration difficulties; 7, Lassitude; 8, Inability to feel; 9, Pessimistic thoughts; 10, Suicidal thoughts. Each item was scored using a scale of 0 to 6 (a higher score indicates increased severity). The maximum total score is 60; 0, no depression; 60, severely depressed. A MADRS remitter is defined as a participant with a MADRS total score <=11 at Week 8.
Time Frame: Week 8
Population: FAS. Missing values were imputed using LOCF.
Measure: Number; unit: participants
Arm/Group | Placebo | 323U66 SR 150 mg | 323U66 SR 300 mg
Number analyzed (Participants) | 186 | 190 | 188
participants | 53 | 60 | 56

6. Secondary Outcome: Number of Clinical Global Impression-Global Improvement (CGI-GI) Responders at Week 8
Description: A CGI-GI assessment was performed at Week 8 (or withdrawal) in comparison with severity in depression observed at Baseline (Week 0; no actual assessment was performed at Baseline [the comparison was subjective]), by using scores from 0 to 7: 0, Not assessed; 1, Very much improved; 2, Much improved; 3, Minimally improved; 4, No change; 5, Minimally worse; 6, Much worse; 7, Very much worse. A CGI-GI responder is defined as a participant with a CGI-GI score of very much improved or much improved at Week 8.
Time Frame: Week 8
Population: FAS. Missing values were imputed using LOCF. Only those participants who were available at Week 8 were analyzed.
Measure: Number; unit: participants
Arm/Group | Placebo | 323U66 SR 150 mg | 323U66 SR 300 mg
Number analyzed (Participants) | 177 | 186 | 173
participants | 100 | 103 | 98

7. Secondary Outcome: Change From Baseline in the Clinical Global Impression-Severity of Illness (CGI-SI) Scores at Weeks 1, 2, 4, 6, and 8
Description: A CGI-SI assessment was performed in terms of severity in depression, by using scores from 0 to 7: 0, Not assessed; 1, Normal, not at all ill; 2, Borderline mentally ill; 3, Mildly ill; 4, Moderately ill; 5, Markedly ill; 6, Severely ill; 7, Among the most extremely ill participants. Change from Baseline in the CGI-SI score was calculated as the value at Week 1, 2, 4, 6, and 8 minus the value at Baseline. The least squared means were estimated based on the ANCOVA model including Baseline CGI-SI score and region as covariates.
Time Frame: Baseline; Weeks 1, 2, 4, 6, and 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | 323U66 SR 150 mg | 323U66 SR 300 mg
Number analyzed (Participants) | 186 | 190 | 188
Scores on a scale
  Week 1, n=182, 187, 184 | -0.2 (0.03) | -0.1 (0.03) | -0.1 (0.03)
  Week 2, n=186, 190, 188 | -0.3 (0.04) | -0.3 (0.04) | -0.2 (0.04)
  Week 4, n=186, 190, 188 | -0.7 (0.06) | -0.5 (0.06) | -0.6 (0.06)
  Week 6, n=186, 190, 188 | -0.9 (0.07) | -0.9 (0.07) | -0.9 (0.07)
  Week 8, n=186, 190, 188 | -1.2 (0.08) | -1.2 (0.08) | -1.1 (0.08)

8. Secondary Outcome: Change From Baseline in the Inventory of Depressive Symptomatology-Self Report (IDS-SR) Total Score at Weeks 1, 2, 4, 6, and 8
Description: The IDS-SR is a 30-item scale used to evaluate the severity and changes in depressive symptoms. Each item was scored from 0 (no symptoms) to 3 (greatest symptom severity). The maximum total score is 84 (0: no symptoms; 84: greatest symptom severity), as participants were asked to answer either item 11 (decreased appetite) or item 12 (increased appetite) (not both) and either item 13 (decreased weight) or item 14 (increased weight) (not both). Change from Baseline was calculated as the value at Week 1, 2, 4, 6, and 8 minus the value at Baseline. The least squared means were estimated based on the ANCOVA model including Baseline IDS-SR score and region as covariates.
Time Frame: Baseline; Weeks 1, 2, 4, 6, and 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | 323U66 SR 150 mg | 323U66 SR 300 mg
Number analyzed (Participants) | 186 | 190 | 188
Scores on a scale
  Week 1, n=182, 187, 184 | -4.8 (0.57) | -4.2 (0.57) | -3.9 (0.57)
  Week 2, n=186, 190, 188 | -6.9 (0.68) | -6.7 (0.68) | -5.8 (0.68)
  Week 4, n=186, 190, 188 | -9.7 (0.82) | -9.3 (0.82) | -8.2 (0.81)
  Week 6, n=186, 190, 188 | -11.5 (0.88) | -12.3 (0.88) | -10.9 (0.87)
  Week 8, n=186, 190, 188 | -13.6 (0.95) | -14.5 (0.95) | -12.6 (0.94)

9. Secondary Outcome: Change From Baseline in the IDS-SR Subscores for Energy, Pleasure, and Interest at Weeks 1, 2, 4, 6, and 8
Description: The IDS-SR is a 30-item scale used to evaluate the severity and changes in depressive symptoms. Each item was scored from 0 (no symptoms) to 3 (greatest symptom severity). Only five items (item 19: general interest; item 20: energy level; item 21: capacity for pleasure or enjoyment, excluding sex; item 22: interest in sex; item 30: leaden paralysis/physical energy) were evaluated for this endpoint, as a subset of the total score. The lowest possible total score and subset total score of IDS-SR are 0 and 0, and the highest possible total score and subset total score of IDS-SR are 84 and 15, respectively. Change from Baseline was calculated as the value at Week 1, 2, 4, 6, and 8 minus the value at Baseline. The least squared means were estimated based on the ANCOVA model including Baseline IDS-SR subscore and region as covariates.
Time Frame: Baseline; Weeks 1, 2, 4, 6, and 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | 323U66 SR 150 mg | 323U66 SR 300 mg
Number analyzed (Participants) | 186 | 190 | 188
Scores on a scale
  Week 1, n=182, 187, 184 | -1.1 (0.16) | -0.9 (0.16) | -0.9 (0.16)
  Week 2, n=186, 190, 188 | -1.3 (0.18) | -1.2 (0.18) | -1.3 (0.18)
  Week 4, n=186, 190, 188 | -2.1 (0.20) | -1.8 (0.20) | -2.0 (0.20)
  Week 6, n=186, 190, 188 | -2.5 (0.22) | -2.6 (0.22) | -2.5 (0.22)
  Week 8, n=186, 190, 188 | -2.9 (0.24) | -3.1 (0.24) | -3.0 (0.24)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of investigational product until the completion of the Follow-up Phase (up to 12 weeks from the start of the Run-in Phase).
Description: SAEs and non-serious AEs were collected in members of the Safety Population, comprised of all participants who took at least one dose of investigational product.
Arm/Group | Placebo | 323U66 SR 150 mg | 323U66 SR 300 mg
Serious Adverse Events (participants affected / at risk) | 2/186 | 2/190 | 1/189
Other Adverse Events (participants affected / at risk) | 63/186 | 62/190 | 80/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=186) | 323U66 SR 150 mg (N=190) | 323U66 SR 300 mg (N=189)
Pyrexia (General disorders) | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=186) | 323U66 SR 150 mg (N=190) | 323U66 SR 300 mg (N=189)
Nasopharyngitis (Infections and infestations) | 35 | 26 | 29
Dry mouth (Gastrointestinal disorders) | 8 | 12 | 28
Headache (Nervous system disorders) | 13 | 15 | 19
Nausea (Gastrointestinal disorders) | 15 | 13 | 16
Constipation (Gastrointestinal disorders) | 3 | 8 | 11
Insomnia (Psychiatric disorders) | 6 | 0 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.